CLINICAL TRIAL: NCT06210269
Title: Oral Antibiotic Outpatient Therapy vs. Placebo in the Treatment of Uncomplicated Acute Appendicitis: a Randomized Double-blind Placebo-controlled Noninferiority Trial APPAC IV
Brief Title: Oral Antibiotic Outpatient Therapy vs. Placebo in the Treatment of Uncomplicated Acute Appendicitis
Acronym: APPAC IV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Oulu University Hospital (Other); Kuopio University Hospital (Other); Pori Central Hospital (Unknown); Jyväskylä Central Hospital (Other); Mikkeli Central Hospital (Other); Seinajoki Central Hospital (Other); Päijänne Tavastia Central Hospital (Other)
Responsible Party: Principal Investigator, Paulina Salminen, Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APPAC IV
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Uncomplicated Acute Appendicitis
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinding. The colored oral capsules for both study groups will have an identical appearance preventing both specific smell and taste; all drugs will be manufactured with identical labelling. Patients randomly assigned to antibiotics will receive oral moxifloxacin 400 mg once daily for seven days. The patients randomly assigned to placebo will receive an identical once daily oral administration and treatment duration of seven days. If the patient is suspected of not responding to the administered treatment based on clinical findings, the patient will undergo laparoscopic appendectomy based on the decision by the surgeon on call and the reasons for proceeding to appendectomy are recorded. Surgical findings and histopathological examination of the removed appendix will be used to confirm the diagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic treatment (Active Comparator): Oral moxifloxacin 400 mg once daily for seven days
  Interventions: Drug: Moxifloxacin 400mg
- Placebo (Active Comparator): Identical oral administration and treatment duration of seven days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Moxifloxacin 400mg — Oral antibiotic
  Arms: Antibiotic treatment
Other: Placebo — Oral placebo
  Arms: Placebo

SUMMARY:
APPAC IV, a randomized double-blind multicenter clinical trial comparing once daily oral moxifloxacin with placebo in an outpatient setting aims to evaluate whether antibiotics and hospitalization or both can be omitted in the treatment of uncomplicated appendicitis further significantly increasing cost savings and patient satisfaction. This is a direct research continuum to the previous trial triad: APPAC, APPAC II and APPAC III, which have already established that the majority of patients with uncomplicated acute appendicitis can be safely treated without surgery. The APPAC IV trial is based on a novel concept and approach to further optimize the nonoperative treatment of uncomplicated acute appendicitis with a high potential in resulting in major health care cost savings and potentially also in significant reduction of antibiotic use in an extremely common surgical emergency.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common surgical emergencies worldwide. For over a century, surgical removal of the appendix has been considered the only possible treatment option with appendectomy still being one of the most common emergency surgeries. Although appendectomy is generally well tolerated, it is a major surgical intervention and can be associated with postoperative morbidity. Since the time Fitz described the relationship between the appendix and pelvic abscess and McBurney demonstrated reduced morbidity from pelvic infections attributable to appendectomy, it has been thought that acute appendicitis invariably progresses to perforation strengthening the belief that emergency appendectomy is always required for acute appendicitis. However, it is now acknowledged that complicated and uncomplicated appendicitis are two different diseases both epidemiologically and clinically also suggesting different pathophysiology and the majority of the cases are uncomplicated. The differential diagnosis is essential as patients presenting with an uncomplicated acute appendicitis may not require surgical intervention and might experience even spontaneous resolution without perforation.

APPAC IV builds on trials by the APPAC (APPendicitis ACuta) study group showing that imaging confirmed uncomplicated acute appendicitis is in fact not a surgical emergency. Antibiotic therapy alone has been shown to be a safe and effective treatment option for patients with computed tomography (CT) confirmed uncomplicated acute appendicitis also in other randomized clinical trials (RCTs). A major knowledge gap on the role of antibiotics still exists. Changing the over century-old dogma of appendectomy for all appendicitis cases into current knowledge where the majority of patients with uncomplicated acute appendicitis can be treated with antibiotics alone if not only with symptomatic therapy, protecting patients from potential adverse effects of antibiotics. In any case, nonoperative treatment, i.e., avoiding unnecessary surgeries will result in major cost and resource savings as the majority of appendicitis cases are uncomplicated. In addition to direct cost savings demonstrated by the APPAC trial at both short- and long-term follow-up, the non-operative treatment approach in this very common surgical emergency allows for the re-allocation of limited health care resources.

Implementing the best available knowledge and current state-of-the-art diagnostics for uncomplicated acute appendicitis using uniform and standardized diagnostic criteria optimizing the pre-intervention patient selection, the investigators anticipate APPAC IV trial to have an even higher success rate of antibiotic treatment for imaging confirmed uncomplicated acute appendicitis compared to the previous trial. Future research should focus on determining both standardized uniform definitions differentiating between appendicitis severity ruling out complicated acute appendicitis and factors predicting non-responsiveness to antibiotics. Further optimizing the patient selection for non-operative treatment would enable potential outpatient management of uncomplicated acute appendicitis resulting in major hospital resource and cost savings. With the current knowledge provided by the landmark APPAC trials and other recent RCTs, initial antibiotic management is consistently associated with a lower complication rate and an at least 70% chance of avoiding surgery within the first year. This information should form the basis of shared informed decision-making.

Aims of the study and study hypothesis

APPAC IV, a randomized double-blind multicenter clinical trial comparing once daily oral moxifloxacin with placebo in an outpatient setting, assesses whether antibiotics and hospitalization or both can be omitted in the treatment of uncomplicated appendicitis further significantly increasing cost savings and patient satisfaction. This is a direct and ambitious research continuum to the previous three APPAC trials, which still have not solved the role and necessity of antibiotics. The APPAC IV is based on a novel concept of symptomatic treatment only further optimizing the possibilities of nonoperative treatment for uncomplicated acute appendicitis. After APPAC IV, it will be known whether antibiotics are needed. Bridging this knowledge gap will lay the foundation for clinical guidelines of nonoperative appendicitis treatment. In any outcome, there is a very high potential of both major health care cost and resource savings. If antibiotics are not needed, this will additionally result in significant reduction of antibiotic use in an extremely common surgical emergency. In addition, as AMR is a major global threat, the APPAC IV trial will include a translational MAPPAC II substudy at TUCH and UTU assessing the effects of antibiotics on gut microbiota, gut health, and correlation to serum cytokines in this real-life randomized patient cohort. As a part of ethical conduct of clinical trials, the investigators will use this unique opportunity of placebo vs. antibiotics randomized patients with the same disease in similar environments to investigate the development of AMR and the underlying bacterial defence mechanisms in Escherichia coli and across the microbiome.

To achieve this, the APPAC IV study including the substudy on microbiology (MAPPAC II) has four specific Aims:

I. Can antibiotics be omitted in the treatment of uncomplicated acute appendicitis? APPAC IV will be a non-inferiority trial with the study hypothesis that oral placebo is noninferior to oral antibiotics in the treatment of CT-confirmed uncomplicated acute appendicitis evaluated at 30 days after the intervention. The primary outcome will be treatment success defined similarly as in the previous APPAC trials in order to enhance comparability and generalizability. This study hypothesis is supported by the APPAC III pilot feasibility trial results where antibiotics were not superior to placebo warranting a large noninferiority trial to truly assess the role of antibiotics in the treatment of uncomplicated acute appendicitis. The expected outcome according to the study hypothesis is that still the majority of patients can be treated without surgery and even antibiotics could perhaps be omitted having a major impact on the antibiotic usage in this very common disease. The successful nonoperative treatment with either antibiotics or symptomatic therapy will in any case result in significant cost savings as almost 60-70% of all appendectomies could be avoided - for example, in the US this would mean approximately almost 200.000 appendectomies and in Europe approximately 550.000 avoided surgeries allowing re-allocation of this major health care resource.

To further improve patient selection and subsequently the success rate of nonoperative treatment for uncomplicated acute appendicitis, accurate differential diagnosis between uncomplicated and complicated acute appendicitis ruling out the former is essential. Potential pre-intervention findings associated with primary non-responsiveness to antibiotics in the APPAC II trial were assessed and appendiceal diameter ≥ 15mm on CT and a body temperature of > 38°C on admission were associated with primary non-responsiveness to antibiotic therapy. For the APPAC IV trial, the additional novel findings of the appendiceal diameter and body temperature have been added to the trial exclusion criteria.

II. Is outpatient treatment of uncomplicated acute appendicitis safe - can hospitalization be avoided? The hospitalization in the previous RCTs was quite long to ensure patient safety. As the current available trials have shown nonoperative treatment to be safe for both oral antibiotics and also for symptomatic therapy in patients with CT-confirmed uncomplicated acute appendicitis, the second aim of APPAC IV trial will be to assess the safety and feasibility of outpatient treatment significantly reducing the need for hospital resources. The patients will be discharged from the emergency room with the oral double-blind medications with no hospital stay unless they are evaluated to require follow-up at the hospital based on the surgeon decision or patient related factors. In order to ensure patient safety, the study coordinator will contact all patients at day 1 after randomization and at 3-4 days together with recommended laboratory tests (leukocyte count and CRP). The hypothesis is that hospitalization in most cases can be avoided having a phenomenal impact on the used health care resources - avoiding hospitalization in most patients will increase the potential high gain and significant impact of the trial in both cost savings, but also allows re-allocation of limited hospital resources.

III. Is there an effect of oral antibiotic treatment on gut microbiota and its antibiotic resistance reservoir (APPAC IV substudy at Turku University hospital: Microbiology APPendicitis Acuta, MAPPAC II) Our initial MAPPAC study has evaluated the differences of appendiceal microbiota between uncomplicated and complicated acute appendicitis showing that these two forms of acute appendicitis have different appendiceal microbiome profiles further supporting the disconnection between these two different forms of acute appendicitis. The aim of the MAPPAC II is to assess the effect of moxifloxacin on gut microbiota in a longitudinal single center prospective cohort study as a part of the APPAC IV clinical trial at the main research center Turku University Hospital. Our hypothesis is that antibiotics will have a notable effect on gut microbiota composition, functional capacity of gut microbiota and its resistome. Effects will be studied from rectal and fecal samples collected both pre- and post-treatment time points by modern, up to date metagenomic shotgun sequencing methodology. Antibiotic resistant bacterial strains by selective bacterial isolation, phenotypic antimicrobial susceptibility testing and whole genome sequencing are studied. Further, the development of antibiotic resistance within gut microbiota will be evaluated in Escherichia coli and across the microbiome using a very recently developed single-cell technology. The investigators will also detect resistance genes from the microbiome with metagenomic sequencing to evaluate the impact of the antibiotic treatment to the whole gut microbiome to show if the results from the E. coli can be extrapolated to the wider community. This will also show if the resistance genes (on plasmids) are from the E. coli population or from other resistant bacteria in the microbiome.

In addition, MAPPAC II will explore the metagenomic data to trace the activity of bacterial CRISPR defense systems in order to address their role in mobile antibiotic resistance.

IV. The effect of oral antibiotic treatment on gut microbiota, development of dysbiosis and related systemic low-grade inflammation and immune response. Gut microbiota correlation to serum cytokine profiles (MAPPAC II).

Cytokines regulate the quantity and quality of inflammatory responses to maintain gut homeostasis. Our recent findings indicate that patients diagnosed with the complicated form of acute appendicitis show a significant increase in several serum cytokines compared with patients diagnosed with the uncomplicated form of appendicitis. This suggests that serum cytokines may serve as diagnostic biomarkers for differentiating uncomplicated and complicated appendicitis. Since antibiotics dramatically change the gut flora and cause at least a transient unbalanced state possibly leading to dysbiosis and systemic low-grade inflammation, we will investigate how serum cytokines and other inflammatory markers and metabolomics profiles are affected by the moxifloxacin treatment, and how this correlates with gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age 18-60 years
3. CT scan confirmed diagnosis of uncomplicated acute appendicitis.

Exclusion Criteria:

1. Complicated acute appendicitis on CT (presence of appendicolith, perforation, abscess, suspicion of tumor, or appendiceal diameter ≥ 15 mm),
2. body temperature > 38°C,
3. age younger than 18 or older than 60 years,
4. contraindications for CT (pregnancy, lactation, allergy to contrast media or iodine, renal insufficiency with serum creatinine exceeding upper reference limit, type 2 diabetes and metformin medication),
5. severe systemic illness (malignancy, or requiring immunosuppressant medication), and
6. all contraindications and other relevant precautions to moxifloxacin (please see list below)
7. inability to co-operate and give informed consent.

Contraindications and other relevant precautions to moxifloxacin in addition to already mentioned trial exclusion criteria: Hypersensitivity to moxifloxacin, or to other quinolones Patients with a history of tendon disease/disorder related to quinolone treatment, Congenital or documented acquired QT prolongation or baseline QTc ≥500 ms, Electrolyte disturbances, particularly in uncorrected hypokalaemia, Clinically relevant bradycardia, Clinically relevant heart failure with reduced left-ventricular ejection fraction, Previous history of symptomatic arrhythmias, Concurrent use of other drugs that prolong the QT interval,

* Anti-arrhythmics class IA (e.g. quinidine, hydroquinidine, disopyramide)
* Anti-arrhythmics class III (e.g. amiodarone, sotalol, dofetilide, ibutilide)
* Antipsychotics (e.g. phenothiazines, pimozide, sertindole, haloperidol, sultopride)
* Tricyclic antidepressive agents
* Certain antimicrobial agents (saquinavir, sparfloxacin, erythromycin IV, pentamidine, antimalarials particularly halofantrine)
* Certain antihistaminics (terfenadine, astemizole, mizolastine)
* Others (cisapride, vincamine IV, bepridil, diphemanil).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 498 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success. | 30 days after treatment initiation
  The primary outcome is 30-day treatment success defined similarly as in the previous trials, i.e. resolution of acute appendicitis resulting in discharge from the hospital without appendectomy during the 30-day follow-up.

SECONDARY OUTCOMES:
Post-intervention complications | 20 years
  Complications according to the Clavien-Dindo classification
Late recurrence of appendicitis | 20 years
  Recurrence of acute appendicitis after the 30-day follow-up.
Hospital stay | 20 years
  Duration of hospital stay in hours
Admission to hospital | 20 years
  Admission to hospital and reason for admission, readmissions to emergency department or hospitalization.
VAS score (visual analogue score) | 20 years
  Pain defined by VAS pain score (scale 0-10, 0 equals no pain and 10 maximum pain imaginable)
Quality of life EQ-5D-5L | 20 years
  Quality of life (QOL, EQ-5D-5L). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Sick leave | 20 years
  Duration of sick leave in days
Treatment costs | 20 years
  Overall treatment and societal costs.
Prognostic factors predicting initial unresponsiveness or recurrent appendicitis | 20 years
  Potential prognostic factors predicting initial unresponsiveness to the randomized treatment as well as recurrent appendicitis
True appendicitis recurrence | 20 years
  True appendicitis recurrence rate following initial successful non-operative treatment as well as the final clinical diagnosis for all operated patients will be evaluated based on the intraoperative and histopathological findings
Subgroup analysis of eligible, not randomized patients | 5 years
  Subgroup analysis of eligible, not randomized patients on all secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, Professor, Principal Investigator — Turku University Hospital Professor of surgery
Locations (9):
- Finland (9):
  - Jyväskylä Central Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Lahti Central Hospital, Lahti
  - Mikkeli Central Hospital, Mikkeli
  - Oulu University Hospital, Oulu
  - Pori Central Hospital, Pori
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Lund H, Haijanen J, Suominen S, Hurme S, Sippola S, Rantanen T, Rautio T, Mattila A, Pinta T, Nordstrom P, Kossi J, Ilves I, Salminen P. A randomized double-blind noninferiority clinical multicenter trial on oral moxifloxacin versus placebo in the outpatient treatment of uncomplicated acute appendicitis: APPAC IV study protocol. Scand J Surg. 2025 Mar;114(1):3-12. doi: 10.1177/14574969241293018. Epub 2024 Dec 5. PMID 39636024